Speech and Brain Research Group (Prof. Kate Watkins) Department of Experimental Psychology University of Oxford

Experimental Psychology



Email: <a href="mailto:speechbrainlab@gmail.com">speechbrainlab@gmail.com</a>

## **PARTICIPANT CONSENT FORM**

CUREC Approval Reference: R52173/RE001 Version 1.0 date 15<sup>th</sup> September 2017

## Investigating non-invasive brain stimulation to enhance fluency in people who stutter (INSTEP)

Purpose of Study: To evaluate speech fluency, brain structure and function in participants who stutter and fluent controls.

| | | Please initial each<br>box |
|---|---|---|
| 1 | I confirm that I have read and understand the information sheet versiondated for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, and without any adverse consequences or academic penalty. | |
| 3 | I understand that research data collected during the study may be looked at by designated individuals from the University of Oxford where it is relevant to my taking part in this study. I give permission for these individuals to access my data. | |
| 4 | I understand that this project has been reviewed by, and received ethics clearance through, the University of Oxford Central University Research Ethics Committee. | |
| 5 | I understand who will have access to personal data provided, how the data will be stored and what will happen to the data at the end of the project. | |
| 6 | I understand how this research will be written up and published. | |
| 7 | I understand how to raise a concern or make a complaint. | |
| 8 | I consent to being audio and video recorded | |
| 9 | I understand that the MRI scans taken in this study are research scans. They are not useful for medical diagnosis, and that scans are not routinely looked at by a doctor. If a concern is raised about a possible abnormality on my scan, I will be informed if a doctor thinks it is medically important. I understand that I would not be informed if the doctor does not think the finding has clear implications for my current or future health. | |
| 10 | I agree to take part in the above study. | |

| Name of r | person taking consent | <br>Date | . <u> </u> |
|---|---|---|---|
| Name of Participant | | Date | Signature |
| | contacting me about futu | · · | |
| Optional: | - | | |
| Optional: | And that this includes research meetings, teaching, and public outreach (please note that you can leave these boxes blank or delete as appropriate if you would prefer us not to use your recordings for these purposes). Please note, also, that we will not give these recordings to individuals outside of the research group. I agree for research data collected in this study to be given to researchers, including those working outside of the EU, to be used in other research studies. I understand that any data that leave the research group will be fully anonymised so that I cannot be identified. Please note that we will not share audio and video recordings. | | |
| Optional: | I agree that the audio an (i.e. training of research s | _ | may be used for educational purposes |

When completed: 1 copy for participant; 1 copy for researcher site file